CLINICAL TRIAL: NCT00905515
Title: Optima: Optimizing Prograf Therapy in Maintenance Allografts II
Acronym: OPTIMAII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Principal Investigator, Paul Bolin, Chair of Internal Medicine, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MR-06-001
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Results first posted 2013-02-11 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Kidney Transplantation
Keywords: Kidney Transplantation; Immunosuppressive Agents
MeSH Terms: interventions — Cyclosporine; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group Cyclosporine (Active Comparator): Maintain on Cyclosporine (CsA) at target trough level of 50-250 ng/mL.
  Interventions: Drug: cyclosporine
- Low Trough Level Prograf Group (Active Comparator): Convert to Prograf (TAC) at target trough levels of 3.0-5.9 ng/mL.
  Interventions: Drug: Prograf (Tacrolimus)
- High Trough Level Prograf Group (Active Comparator): Convert to TAC at target trough levels of 6.0-8.9 ng/mL.
  Interventions: Drug: Prograf (Tacrolimus)

INTERVENTIONS:
Drug: cyclosporine — Maintain on cyclosporine at target trough level of 50-250 ng/mL.
  Other Names: Cyclosporine/Neoral®/Sandimmune®/Gengraf®
  Arms: Control Group Cyclosporine
Drug: Prograf (Tacrolimus) — Convert to Prograf at target trough levels of 3.0-5.9 ng/mL (Arm 2) or target trough levels of 6.0-8.9 ng/mL (Arm 3).
  Other Names: Tacrolimus/Prograf®/FK506
  Arms: High Trough Level Prograf Group; Low Trough Level Prograf Group

SUMMARY:
This study is designed to optimize calcineurin immunosuppressive regimens and evaluate immunological and non-immunological markers that may explain mechanistic differences in these agents and their effects.

DETAILED DESCRIPTION:
One of the major challenges in transplantation over the past two decades has been managing long-term renal function. Serum creatinine is the most commonly used serum marker of renal function. However serum creatinine is insensitive for detecting small decreases in glomerular filtration rate (GFR). Another marker for renal function is cystatin C. Dharnidharka et al concluded that cystatin C is superior to serum creatinine as a marker of kidney function since cystatin C was a more sensitive marker than serum creatinine for detecting decreases in GFR. Pirsch et al reported that tacrolimus-treated patients had a lower incidence of severe acute rejection and better lipid profiles than cyclosporine-treated patients.

Cardiovascular disease is the primary cause of premature death in renal and other transplant recipients. Current immunosuppressive protocols often elevate cardiovascular disease risk factors such as hypertension, hyperlipidemia, obesity and diabetes.

This study is designed to optimize calcineurin immunosuppressive regimens to ensure the best possible long-term outcomes after renal transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient is the recipient of a cadervic or living donor renal transplant.
* Patient was 18 years of age at time of transplant.
* Patient is at least 6 months post-transplant.
* Patient has been on a cyclosporine-based immunosuppressive regimen since the transplant.
* Patient has a functioning allograft and a Cockcroft/Gault estimate of creatinine clearance >or= 35 mL/min within four weeks prior to randomization.
* Patient or legal guardian has signed and dated an Institutional Review Board (IRB) approved informed consent document and is willing and able to follow study procedures.
* Females are not pregnant and agree to practice effective birth control while receiving immunosuppressant medication.

Exclusion Criteria:

* Patient is the recipient of a solid organ transplant other than the kidney.
* Patient experienced biopsy-confirmed, acute rejection, (Banff 97 criteria)within 3 months before randomization that required treatment, which is defined as antilymphocyte therapy, corticosteroids, or an increase in the number or dose of immunosuppressant medication.
* Patient has recurrence of primary renal disease, or de novo renal disease.
* Patient has a urine protein of > 1.5g/24 hours or two successive urinalyses sent to and reported by the laboratory indicating albuminuria greater than 2+ within 6 months prior to enrollment.
* Patient has an estimated creatinine clearance < 35 mL/min calculated using Cockcroft/Gault formula within four weeks prior to randomization.
* Patient has changed adjunctive immunosuppressant therapy within one month if randomization.
* Patient is pregnant or lactating.
* Patient is a known carrier of any of the HIV viruses.
* Patient has a known or suspected malignancy (except for treated squamous or basal cell skin cancers) < 5 years before randomization or a history of post-transplant lymphoproliferative disease (PTLD).
* Patient has a known hypersensitivity to tacrolimus, or any of the excipients of the drug.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2003-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bolin, MD, Principal Investigator — East Carolina University
Locations (1):
- Brody School of Medicine at East Carolina University, Greenville, North Carolina, United States

REFERENCES:
- [Background] Dharnidharka VR, Kwon C, Stevens G. Serum cystatin C is superior to serum creatinine as a marker of kidney function: a meta-analysis. Am J Kidney Dis. 2002 Aug;40(2):221-6. doi: 10.1053/ajkd.2002.34487. PMID 12148093
- [Background] Pirsch JD, Miller J, Deierhoi MH, Vincenti F, Filo RS. A comparison of tacrolimus (FK506) and cyclosporine for immunosuppression after cadaveric renal transplantation. FK506 Kidney Transplant Study Group. Transplantation. 1997 Apr 15;63(7):977-83. doi: 10.1097/00007890-199704150-00013. PMID 9112351

RESULTS

PARTICIPANT FLOW:
Groups:
- Remaining on CsA: Stable transplant recipients randomly assigned to continue on Cyclosporine (CsA( with a target trough level of 50-250 ng/mL.
- Reduced TAC: Stable transplant recipients randomly assigned to convert to "reduced" Tacrolimus (TAC) with target trough levels 3.0-5.9 ng/mL.
- Standard TAC: Stable transplant recipients randomly assigned to convert to "standard" TAC with target trough levels of 6.0-8.9 ng/mL.
Period: Overall Study
Arm/Group | Remaining on CsA | Reduced TAC | Standard TAC
Started | 21 | 20 | 22
Completed | 19 | 20 | 20
Not Completed | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Remaining on CsA: Patients remained on CSA and were not converted to TAC.
- Reduced TAC: Patients converted from CsA to TAC with trough concentrations 3.0-5.9 ng/mL
- Standard TAC: Patients were converted from CsA to TAC with trough concentrations of 6.0-8.9 ng/mL
- Total: Total of all reporting groups
Arm/Group | Remaining on CsA | Reduced TAC | Standard TAC | Total
Number analyzed (Participants) | 21 | 20 | 22 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 16 | 14 | 43
  >=65 years | 8 | 4 | 8 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.65 (12.036) | 58.57 (12.023) | 59.14 (10.011) | 58.48 (11.196)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 3 | 19
  Male | 15 | 10 | 19 | 44
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 22 | 63

OUTCOME MEASURES:

1. Primary Outcome: Renal Function in Patients Converted From Cyclosporine to Prograf
Time Frame: 3 years
Measure: Mean (Full Range); unit: Change in serum creatinine (mg/dL)
Groups:
- Remaining on CsA: Stable transplant recipients randomly assigned to continue on CSA with a target trough level of 50-250 ng/mL.
- Reduced TAC: Stable transplant recipients randomly assigned to convert to "reduced" TAC with target trough levels 3.0-5.9 ng/mL.
Arm/Group | Remaining on CsA | Reduced TAC | Standard TAC
Number analyzed (Participants) | 21 | 20 | 22
Change in serum creatinine (mg/dL) | 0.05 [-0.04 to 0.14] | 0 [0 to 0] | 0.10 [-0.07 to 0.26]

2. Primary Outcome: Optimal Dose of Calcineurin Inhibitor in Long-term Maintenance Kidney Transplant Patients
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Remaining on CsA | Reduced TAC | Standard TAC
Number analyzed (Participants) | 21 | 20 | 22
ng/dL | 130.2 (54.94) | 5.24 (2.06) | 6.90 (2.06)

3. Primary Outcome: Change in Risk Factors for Cardiovascular Morbidity and Chronic Graft Dysfunction as Evidenced by Blood Levels of Homocysteine
Time Frame: 3 years
Measure: Median (Standard Deviation); unit: ng/dL
Arm/Group | Remaining on CsA | Reduced TAC | Standard TAC
Number analyzed (Participants) | 21 | 20 | 22
ng/dL | 4.75 (0.82) | 4.72 (0.52) | 4.89 (0.33)

ADVERSE EVENTS:
Arm/Group | Remaining on CsA | Reduced TAC | Standard TAC
Serious Adverse Events (participants affected / at risk) | 0/21 | 2/20 | 1/22
Other Adverse Events (participants affected / at risk) | 11/21 | 14/20 | 14/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remaining on CsA (N=21) | Reduced TAC (N=20) | Standard TAC (N=22)
New onset diabetes mellitus (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remaining on CsA (N=21) | Reduced TAC (N=20) | Standard TAC (N=22)
Bone Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Blood Glucose (Endocrine disorders) | 7 (12) | 9 (23) | 8 (17)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Gingival Hypertrophy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Absolute Neutrophil (Blood and lymphatic system disorders) | 1 (1) | 10 (11) | 10 (10)
Hirsutism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No